CLINICAL TRIAL: NCT02687737
Title: Genioglossus Motor Recruitment During Swallowing and Expiratory Loading Exercises
Brief Title: Tongue Motor Recruitment During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201600120
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Tongue; Genioglossus; genioglossus recruitment
MeSH Terms: interventions — Neurofeedback; Barium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental): The participants will have the following tests performed: Maximum Expiratory Pressure (MEP), insertion of a fine-wire electromyography (EMG) electrode into the mid-line base of the tongue, will complete swallowing tasks and breathing tasks under Videofluoroscopy (fluoroscopy on only during the actual task)
  Interventions: Procedure: Electromyography; Procedure: Maximum expiratory pressure; Procedure: Videofluoroscopy; Behavioral: Swallowing Tasks

INTERVENTIONS:
Procedure: Electromyography — During the fine wire electromyography (EMG), the participant will be asked to complete breathing exercises at 50% and 75% of their maximum capacity (determined prior to fine wire EMG using manometry) to determine activation and recruitment of genioglossus muscle.
  Other Names: EMG
Procedure: Maximum expiratory pressure — The participants' maximum expiratory pressure (MEP) will be assessed using a hand-held digital manometer (MP01, Micro Direct Inc.). The subject will be standing and while wearing a nose clip be asked to blow out as hard and fast as they can to determine their MEP. This will be completed a maximum of three times to obtain values within close range of one another.
  Other Names: MEP
Procedure: Videofluoroscopy — Videofluoroscopy allows for time-synced, frame-by-frame data analysis for the specific measures taken during swallowing tasks.
  Other Names: Videofluoroscopy and Barium
Behavioral: Swallowing Tasks — These include: an anterior tongue press to the alveolar ridge (behind the front molars), a saliva swallow, a 10 mL barium swallow, a 10 mL barium "hard" swallow (i.e. swallowing with extra effort), and two breathing exercise trials at 50% MEP and 75% MEP.

SUMMARY:
The prevalence of dysphagia may be as high as 22% in individuals over 50 years of age. There are few therapeutic options offered to these individuals. One more recent therapeutic option is Expiratory Muscle Strength Training (EMST), which has been used successfully to maintain or increase expiratory force generating pressures, cough function, and swallowing in a number of disease populations. Recently, the investigators have noted improvements in oral transit time during swallowing in individuals with Amyotrophic Lateral Sclerosis (ALS) that could potentially be attributed to improved base of tongue functioning and muscle activation.

There has been one study that demonstrated that breathing training resulted in increased and prolonged submental (under the chin) muscle activation as evidenced by surface electromyography. However, no studies have investigated the activation of the tongue muscles during various swallowing and breathing exercises. A small needle electrode (fine wire EMG) is standard of care in diagnosing muscular diseases because it can determine amount of muscle recruitment for muscles throughout the body. This aim of this research study is to examine the effects of breathing exercises and swallowing exercises on tongue muscle activity in healthy adults.

DETAILED DESCRIPTION:
This study will measure tongue muscle activation using fine wire EMG placed into the tongue muscle (underneath the chin) during swallowing and breathing exercises. A neurologist trained in EMG will perform all procedures to ensure best placement and minimize discomfort of the participant. While the needle is in place, the participant will complete a series of swallowing tasks and breathing exercises using a small, handheld training device. All swallowing and breathing tasks will be viewed under x-ray in order to see the movement and timing of the tongue and swallowing muscles during each task. Participation in the study will take one, one-hour visit to the Shands Dental Tower lab spaces where all procedures will be completed.

ELIGIBILITY:
Inclusion Criteria:

* No known major disease, disorder or medical conditions

Exclusion Criteria:

* Currently on anticoagulant therapy
* Has a bleeding/anticoagulant disorder or disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) will be used to analyze genioglossus muscle movement | Baseline
  Electromyography (EMG) activity will be recorded via standard concentric needle electrodes inserted into the genioglossus muscle. Maximum muscle activation will be recorded and analyzed to determine difference between tasks using the genioglossus muscle.
Kinematic Swallowing Measurements will be used to analyze a normal movement of swallowing | Baseline
  Kinematic swallowing measurements is an objective analysis of videofluoroscopy. This involves capturing and manipulating digital images with computer technology to make exact timing measures of bolus flow and movement of structures, as well as spatial measurements of distance and area against reference points.

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Plowman, PhD, CCC-SLP, Principal Investigator — University of Florida College of Public Health and Health Professions
Locations (1):
- Shands Hospital at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wheeler-Hegland KM, Rosenbek JC, Sapienza CM. Submental sEMG and hyoid movement during Mendelsohn maneuver, effortful swallow, and expiratory muscle strength training. J Speech Lang Hear Res. 2008 Oct;51(5):1072-87. doi: 10.1044/1092-4388(2008/07-0016). Epub 2008 Aug 26. PMID 18728114
- [Background] Trinder J, Woods M, Nicholas CL, Chan JK, Jordan AS, Semmler JG. Motor unit activity in upper airway muscles genioglossus and tensor palatini. Respir Physiol Neurobiol. 2013 Sep 15;188(3):362-9. doi: 10.1016/j.resp.2013.06.011. Epub 2013 Jun 21. PMID 23797183